CLINICAL TRIAL: NCT04522921
Title: Childhood Obesity - Prevention of Diabetes Through Changed Eating Patterns (The COPE-study) - An Non-randomized Intervention Trial Investigating the Efficacy of Dietary Changes in Protein
Brief Title: Childhood Obesity - Prevention of Diabetes Through Changed Eating Patterns
Acronym: COPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: The COPE-study
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-02

CONDITIONS: Childhood Obesity; Overweight and Obesity; Adolescent Obesity; Adolescent Overweight; Diabetes
Keywords: Eating Behavior; Eating Habit; Quality of Life; Dietary Habits; Eating Disorders
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Diabetes Mellitus; Feeding Behavior; Feeding and Eating Disorders | interventions — Diet; Methods

STUDY DESIGN:
Intervention Model Description: 1. SARS CoV group (former control group): Current weight-loss diet (15E%/day protein) for the 10 weeks they attend the camp, however, due to a COVID19 lockdown of the camps, these children were sent home for five weeks, and therefore excluded from longitudinal comparison between the groups.
  2. Control group (CG): Current weight-loss diet (15E%/day protein) for the 10 weeks they attend the camp.
  2) Intervention group (IG): A higher protein diet (25E%/day) for the 10 weeks they attend the camp.
Who Masked: Participant, Investigator
Masking Description: At enrollment the participants have no knowledge of which group they are assigned.
  The investigator has no knowledge of or influence on how participants are divided into different groups. Participants are assigned groups by the camp staff.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SARS CoV-group (Other): This group should have been the control group. However, due to the COVID19 lockdown of the camps for 5 five weeks, with no control of diet and physical activity, this group could not act as control group. Therefore, this group has been excluded from longitudinal analyses.
  Interventions: Dietary Supplement: Diet with a lower amount of protein (15E% per day)
- Control Group (CG) (Active Comparator): Current weight-loss diet (15E%/day protein) for the 10 weeks they attend the camp. Increased follow-up contact after camp.
  Interventions: Behavioral: Increased follow-up contact after the 10-week intervention; Dietary Supplement: Diet with a lower amount of protein (15E% per day)
- Intervention group (IG) (Experimental): A higher protein diet (25E%/day) for the 10 weeks they attend the camp. Increased follow-up contact after camp.
  Interventions: Dietary Supplement: Diet with a higher amount of protein (25E% per day); Behavioral: Increased follow-up contact after the 10-week intervention

INTERVENTIONS:
Dietary Supplement: Diet with a higher amount of protein (25E% per day) — In a caloric restricted and increased physical activity setting, the participants will be served a higher protein (25E%/day) diet.
  Arms: Intervention group (IG)
Behavioral: Increased follow-up contact after the 10-week intervention — Both the control-group and the intervention-group were offered an increased follow-up contact after camp.
  Arms: Control Group (CG); Intervention group (IG)
Dietary Supplement: Diet with a lower amount of protein (15E% per day) — In a caloric restricted and increased physical activity setting, the participants will be served a low-moderate protein (15E%/day) diet.
  Arms: Control Group (CG); SARS CoV-group

SUMMARY:
The main purpose of the present study is to perform a 10 weeks dietary intervention study with a follow-up for 52 weeks in children from 7-14 years of age with overweight or obesity. In a caloric restricted and increased physical activity setting the control group will consume a low-moderate protein (15E%/day) diet whereas the intervention group will consume a higher protein (25E%/day) diet. Secondary, the investigators want to investigate the effect of frequent follow-up after the intervention, and the overall effect of the lifestyle camp.

Compared to the low-moderate protein diet, the investigators hypothesis that a diet with higher consumption of protein-containing foods will more effectively induce weight loss (a reduction in BMI-SDS) or weight maintenance in children with overweight or obesity, and improve quality of life, and risk factors for type 2 diabetes.

DETAILED DESCRIPTION:
The study will be performed in collaboration with the staff of the well-established multi-component-overnight camps (Julemærkehjem) in Denmark. The multi-component-overnight camps are intensive weight loss camps to which Danish schoolchildren, from 7-14 years of age, are referred to for 10-weeks intervention focusing on healthy lifestyle, healthy eating, new habits and increased physical activity.

The primary outcome is anthropometry (BMI-SDS, fat mass, fat-free mass). Secondary outcomes are metabolic health and questionnaires investigating quality of life, eating behavior traits, eating habits and eating-related problems i.e., overeating and loss of control eating.

The children will be measured at baseline, 10-weeks and at a 52-weeks follow-up visit.

Furthermore, participants will be invited to follow-up visits 3 years, 5 years, 7 years and 10 years, respectively.

ELIGIBILITY:
Inclusion Criteria:

* The child attends a multi-component-overnight camp in Hobro or Fjordmark between October 2020 and March 2022.
* The child is between 7 and 14 years of age (inclusive) while attending camp.
* At least one parent/guardian submit written and oral consent to participate with his/her child.
* Parent/legal guardian has submitted oral and written consent to participation of their child. In case of shared custody both parents must submit written and oral consent before their child can participate in the trial.

Exclusion Criteria:

* The child has a disease, diagnose or eating disorder that require treatment.
* The child or parent/guardian participate in another clinical trial or plan to do so in the near future.
* The parent/guardian do not understand the written informed consent.
* The child or parent/guardian are unwilling to or unable to comply with the study protocol and instruction given by the study staff.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 211 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2032-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Bruun, Professor, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Weight Loss Camp Hobro, Hobro
  - Weight Loss Camp Fjordmark, Kruså

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jakobsen DD, Brader L, Bruun JM. Effect of a higher protein diet and lifestyle camp intervention on childhood obesity (The COPE study): results from a nonrandomized controlled trail with 52-weeks follow-up. Eur J Nutr. 2024 Sep;63(6):2173-2184. doi: 10.1007/s00394-024-03420-z. Epub 2024 May 9. PMID 38724826
- [Result] Jakobsen DD, Jarvholm K, Brader L, Bruun JM. Long-term changes in eating-related problems and quality of life in children with overweight and obesity attending a 10-week lifestyle camp. Obes Res Clin Pract. 2024 May-Jun;18(3):209-215. doi: 10.1016/j.orcp.2024.04.002. Epub 2024 May 4. PMID 38705820
- [Result] Pauls DD, Clausen L, Bruun JM. Eating behavior profiles in children following a 10-week lifestyle camp due to overweight/obesity and low quality of life: A latent profile analysis on eating behavior. Eat Behav. 2025 Apr;57:101971. doi: 10.1016/j.eatbeh.2025.101971. Epub 2025 Mar 24. PMID 40157300
- [Result] Aagaard I, Jakobsen DD, Bruun JM. Association between quality of life and emotional overeating - a cross-sectional study in Danish children attending a multicomponent lifestyle camp. Eur J Pediatr. 2023 Dec;182(12):5493-5499. doi: 10.1007/s00431-023-05206-7. Epub 2023 Sep 30. PMID 37777600
- [Result] Orry S, Dalstrup Jakobsen D, Kristensen NM, Meldgaard Bruun J. Uric acid and sCD163 as biomarkers for metabolic dysfunction and MAFLD in children and adolescents with overweight and obesity. J Pediatr Endocrinol Metab. 2023 Jun 8;36(7):643-649. doi: 10.1515/jpem-2023-0228. Print 2023 Jul 26. PMID 37285233

RESULTS

PARTICIPANT FLOW:
Groups:
- Control-group (CG): Standard weight-loss diet (15E%/day protein) for the 10 weeks they attend the camp and increased follow-up.
  Increased follow-up contact after attending a weight loss camp: After leaving the camp, the children and their families with increased follow-up contact will be contacted once every month within the first 6 month and once every other month until 52-weeks follow-up (8 times total). The children and their families will be contacted by phone, facetime or skype as they prefer, within a predetermined and known timeframe. The conversation will focus on individual topics chosen by the child/parent.
- Intervention Group (IG): A higher protein diet (25E%/day) for the 10 weeks they attend the camp and increased follow-up.
  Increased follow-up contact after attending a weight loss camp: After leaving the camp, the children and their families with increased follow-up contact will be contacted once every month within the first 6 month and once every other month until 52-weeks follow-up (8 times total). The children and their families will be contacted by phone, facetime or skype as they prefer, within a predetermined and known timeframe. The conversation will focus on individual topics chosen by the child/parent.
- SARS CoV-group: Standard weight-loss diet (15E% of protein) during the camp. However, they were sent home for five weeks due to a COVID19 lockdown.
Period: Overall Study
Arm/Group | Control-group (CG) | Intervention Group (IG) | SARS CoV-group
Started | 75 | 86 | 34
Completed (Participants who completed the 10-week camp intervention including the assigned dietary intervention.) | 71 | 74 | 34 (All participants in this group were excluded from analysis due to a COVID19 lockdown of the camps.)
Not Completed | 4 | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control-group: In the control group, no changes were. This group received a standard care lifestyle camp for 10-weeks.
- Intervention-group: In the intervention group, the aim was to replace carbohydrates-rich foods at breakfast and two in-between meals with naturally protein-containing foods (e.g., dairy products, nuts, egg, meat-products) to increase the amount of protein from ~ 10-15E% to ~ 25E% per day with minimal changes in total caloric intake.
- SARS CoV-group: The SARS CoV-group were affected by the COVID-19 lockdown of the camps.Thus, they were sent home for five weeks with no control of dietary intake and physical activity. They received standard care during their stay at camp.
- Total: Total of all reporting groups
Arm/Group | Control-group | Intervention-group | SARS CoV-group | Total
Number analyzed (Participants) | 75 | 86 | 34 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (1.4) | 12.1 (1.5) | 12.5 (1.1) | 12.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 19 | 90
  Male | 39 | 51 | 15 | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body weight [Mean (Standard Deviation); unit: Kg] | 73.6 (14.6) | 72.7 (18.0) | 73.4 (12.5) | 73.2 (16.5)
Height [Mean (Standard Deviation); unit: Meter] | 1.59 (0.1) | 1.59 (0.1) | 1.60 (0.1) | 1.59 (0.1)
Body mass index standard deviation score (BMI-SDS) [Mean (Standard Deviation); unit: standard deviation] — BMI-SDS is and age-and-sex adjusted BMI score. It was calculated using World Health Organization Anthro-Plus software. A BMI-SDS > 1SD is defined as overweight, and a BMI-SDS> 2SD is defined as obesity.
  standard deviation | 2.65 (0.7) | 2.66 (0.7) | 2.57 (0.6) | 2.65 (0.7)
Body fat [Mean (Standard Deviation); unit: percentage of body fat] — Population: Some participants had missing values on body composition.
  percentage of body fat
    number analyzed (Participants) | 67 | 84 | 34 | 185
    (all) | 41.4 (6.6) | 41.0 (6.8) | 42.4 (6.0) | 41.2 (6.7)
Skeletal muscle mass [Mean (Standard Deviation); unit: Kg] — Population: Some participants had missing values on body composition.
  Kg
    number analyzed (Participants) | 67 | 84 | 34 | 185
    (all) | 23.0 (4.8) | 23.2 (5.8) | 22.8 (4.2) | 23.1 (5.4)
Blood pressure (systolic) [Mean (Standard Deviation); unit: mmHg] — Population: Missing data due to refusal of blood pressure measurements or malfunction of the blood pressure device.
  mmHg
    number analyzed (Participants) | 73 | 68 | 23 | 164
    (all) | 111.1 (10.7) | 109.8 (10.31) | 109.2 (9.1) | 110.5 (10.5)
Blood pressure (diastolic) [Mean (Standard Deviation); unit: mmHg] — Population: Missing data due to refusal of blood pressure measurements or malfunction of the blood pressure device.
  mmHg
    number analyzed (Participants) | 73 | 68 | 23 | 164
    (all) | 70.2 (6.4) | 72.5 (8.7) | 71.7 (5.1) | 71.3 (7.7)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 3.9 (0.7) | 4.3 (0.7) | 4.0 (0.8) | 4.2 (0.7)
HDL cholesterol [Mean (Standard Deviation); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 1.2 (0.3) | 1.2 (0.2) | 1.2 (0.3) | 1.2 (0.2)
LDL cholesterol [Mean (Standard Deviation); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 40 | 11 | 84
    (all) | 2.2 (0.6) | 2.5 (0.6) | 2.2 (0.6) | 2.4 (0.6)
Triglyceride [Median (Inter-Quartile Range); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 1.3 [0.9 to 1.5] | 1.3 [0.9 to 1.8] | 1.3 [0.8 to 1.6] | 1.3 [0.9 to 1.8]
ALAT [Median (Inter-Quartile Range); unit: units/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  units/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 22 [18 to 27] | 22.5 [18 to 33] | 20 [15 to 22] | 22 [18 to 30]
ASAT [Median (Inter-Quartile Range); unit: units/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  units/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 24 [20 to 25] | 23 [20 to 29] | 16 [15 to 23] | 23 [20 to 27]
GGT [Median (Inter-Quartile Range); unit: units/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  units/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 16 [14 to 19] | 16 [13 to 19] | 15 [11 to 19] | 16 [13 to 19]
Basic phosphatase [Mean (Standard Deviation); unit: units/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  units/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 297 (84) | 274 (90) | 251 (77) | 284 (87)
P-glucose [Mean (Standard Deviation); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 5.9 (0.4) | 5.9 (0.3) | 5.9 (0.4) | 5.9 (0.3)
Albumin [Mean (Standard Deviation); unit: g/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  g/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 42.0 (2.4) | 42.8 (2.4) | 43 (1.9) | 42.4 (2.4)
CD163 [Median (Inter-Quartile Range); unit: mg/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mg/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 2.4 [2.0 to 3.1] | 2.6 [2.1 to 3.0] | 2.1 [2.0 to 3.2] | 2.5 [2.0 to 3.1]
Platelets [Mean (Standard Deviation); unit: units/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  units/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 314 (64) | 310 (61) | 295 (29) | 312 (62)
Uric acid [Mean (Standard Deviation); unit: mmol/L] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/L
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 0.31 (0.0) | 0.32 (0.1) | 0.33 (0.1) | 0.31 (0.1)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] — Population: Blood samples were voluntary for all participants; therefore, only a subsample of participants had blood samples collected.
  mmol/mol
    number analyzed (Participants) | 33 | 44 | 11 | 88
    (all) | 34.9 (2.5) | 35.0 (2.1) | 35 (2.8) | 34.9 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index Standard Deviation Score (BMI-SDS)
Description: BMI-SDS was calculated using World Health Organization Anthro-Plus software.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: The COVID-19 pandemic forced a lockdown from December 2020 to February 2021. All children affected by the COVID-19 lockdown (The SARS CoV-group) were sent home for five weeks with no control of dietary intake and physical. Only a subsample of participants had bloodsamples collected.
Measure: Mean (95% Confidence Interval); unit: Standard deviation score
Groups:
- Control Group: In the control group, no changes were. This group received a standard care lifestyle camp for 10-weeks.
- Intervention Group: In the intervention group, the aim was to replace carbohydrates-rich foods at breakfast and two in-between meals with naturally protein-containing foods (e.g., dairy products, nuts, egg, meat-products) to increase the amount of protein from ~ 10-15E% to ~ 25E% per day with minimal changes in total caloric intake.
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 34
Standard deviation score | -0.54 [-0.63 to -0.45] | -0.61 [-0.68 to -0.53] | -0.70 [-0.84 to -0.55]

2. Primary Outcome: Body Weight (kg)
Description: Body weight (kg) was measured in light clothing without shoes using a Bioelectric impedance (InBody model 270, Hopkins Medical Products, Grand Rapids, MI, USA).
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kilogram
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 34
kilogram | -6.25 [-7.54 to -4.96] | -6.62 [-7.87 to -5.37] | -7.64 [-9.47 to -5.81]

3. Primary Outcome: Body Fat (%)
Description: Body fat (%) was measured in light clothing without shoes using a Bioelectric impedance (InBody model 270, Hopkins Medical Products, Grand Rapids, MI, USA).
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage (%)
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 34
Percentage (%) | -5.77 [-6.94 to -4.60] | -6.06 [-7.14 to -4.99] | -7.44 [-9.35 to -5.53]

4. Primary Outcome: Skeletal Muscle Mass (kg)
Description: Skeletal muscle mass (kg) was measured in light clothing without shoes using a Bioelectric impedance (InBody model 270, Hopkins Medical Products, Grand Rapids, MI, USA).
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Kilogram
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 34
Kilogram | 0.22 [-0.17 to 0.61] | -0.003 [-0.42 to 0.41] | 0.49 [-0.10 to 1.09]

5. Secondary Outcome: Body Height (m)
Description: Height (m) was measured using a fixed wall measuring tape.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Meter
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 34
Meter | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.02] | 0.02 [0.01 to 0.03]

6. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured with the right arm placed at heart level using an automatic non-invasive blood pressure monitor (Omron M3, Kyoto, Japan).
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 32
mmHg | -4.39 [-6.68 to -2.09] | -3.32 [-5.97 to -0.67] | -4.38 [-8.53 to -0.23]

7. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 6
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 71 | 74 | 32
mmHg | -2.97 [-4.50 to -1.43] | -4.28 [-6.42 to -2.13] | -5.24 [-8.36 to -2.11]

8. Secondary Outcome: P-cholesterol
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.39 [-0.58 to -0.21] | -0.55 [-0.75 to -0.35] | -0.63 [-0.90 to -0.35]

9. Secondary Outcome: HDL Cholesterol
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.03 [-0.09 to 0.04] | -0.04 [-0.11 to 0.02] | -0.10 [-0.23 to 0.03]

10. Secondary Outcome: LDL Cholesterol
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.25 [-0.42 to -0.09] | -0.43 [-0.60 to -0.26] | -0.34 [-0.56 to -0.12]

11. Secondary Outcome: P-tryglyceride
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.18 [-0.35 to -0.01] | -0.20 [-0.37 to -0.03] | -0.35 [-0.65 to -0.05]

12. Secondary Outcome: ALAT
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
units/L | -0.14 [-0.25 to -0.03] | -0.28 [-0.43 to -0.13] | 0.13 [-0.10 to 0.37]

13. Secondary Outcome: ASAT
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
units/L | -0.04 [-0.14 to 0.06] | -0.16 [-0.27 to -0.04] | 0.18 [0.06 to 0.29]

14. Secondary Outcome: GGT
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
units/L | -0.16 [-0.25 to -0.07] | -0.22 [-0.36 to -0.09] | -0.24 [-0.38 to -0.10]

15. Secondary Outcome: Basic Phosphatase
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
units/L | -15.47 [-36.22 to 5.29] | -3.69 [-25.26 to 17.88] | -22.62 [-45.46 to 0.23]

16. Secondary Outcome: HbA1c
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/mol
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/mol | -0.46 [-1.24 to 0.31] | -0.21 [-0.82 to 0.41] | -0.23 [-0.97 to 0.51]

17. Secondary Outcome: P-glucose
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.07 [-0.18 to 0.04] | -0.02 [-0.11 to 0.07] | -0.01 [-0.12 to 0.09]

18. Secondary Outcome: Albumin
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: g/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
g/L | -0.51 [-1.29 to 0.26] | -0.14 [-0.94 to 0.66] | -2.33 [-3.37 to -1.29]

19. Secondary Outcome: CD163
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mg/L | 0.01 [-0.08 to 0.09] | -0.08 [-0.17 to 0.01] | -0.12 [-0.24 to 0.01]

20. Secondary Outcome: Platelets
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: The COVID-19 pandemic forced a lockdown from December 2020 to February 2021. All children affected by the COVID-19 lockdown (The SARS CoV-group) were sent home for five weeks with no control of dietary intake and physical. Only a subsample of participants had bloodsamples collected. .
Measure: Mean (95% Confidence Interval); unit: Units/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
Units/L | -0.14 [-0.18 to -0.10] | -0.10 [-0.14 to -0.06] | -0.14 [-0.21 to -0.06]

21. Secondary Outcome: Uric Acid
Description: Educated bio-analysts were responsible for collecting blood samples in a subsample of children.
Time Frame: Mean changes from baseline to 10-weeks (post camp intervention)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control Group | Intervention Group | SARS CoV-group
Number analyzed (Participants) | 33 | 42 | 11
mmol/L | -0.04 [-0.05 to -0.02] | -0.03 [-0.04 to -0.02] | -0.02 [-0.05 to 0.007]

ADVERSE EVENTS:
Time Frame: 10-weeks
Description: Since this was a short-term dietary intervention in children, all-cause mortality/adverse events were not systematically monitored. An annual safety report has been submitted to the ethical committee to report any serious side effects, incidents or adverse events. The most recent report, submitted in 2024, indicated that no serious side effects, incidents, or adverse events were reported in any study arm. Therefore, adverse events are reported for all participants across combined arms/groups.
Groups:
- All Arms: As per the annual requirement from the ethics committee, we report side effects, incidents, and adverse events each year. The most recent report, submitted in 2024, indicated that no serious side effects, incidents, or adverse events were reported in any study arm. Therefore the Arms/Groups are pooled in the reporting.
Arm/Group | All Arms
All-Cause Mortality (participants affected / at risk) | 0/195
Serious Adverse Events (participants affected / at risk) | 0/195
Other Adverse Events (participants affected / at risk) | 0/195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT04522921/Prot_SAP_000.pdf